CLINICAL TRIAL: NCT05570136
Title: The Effect of Functional Exercise Interventions for Older Adults With Sarcopenia: A Hybrid Approach Study Aiming for Community Implementation
Brief Title: Functional Exercise for Sarcopenia
Acronym: STEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yi-Ling Hu, Assistant Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202201076B0
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Sarcopenia
Keywords: habit; community; older adult; functional exercise
MeSH Terms: conditions — Sarcopenia; Habits | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The treatment group will receive functional exercise intervention, and the sham control group will receive weekly newsletters and phone calls.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Participants in the treatment group will receive the 12-week STEP by a trained interventionist. In the first four weeks, the interventionist will focus on building participants' selfefficacy and health literacy and help participants learn the STEP exercise and principles. In the following four weeks, the interventionist will help the older adults to be more independent in prescribing exercise activities for themselves. In the last four weeks, participants will be fulling knowledgeable and independent on functional exercising; the interventionist will allocate community resources for long-term maintenance. After program completion, trained raters will administer at post-tests. There will also be a 3-month and 6-month follow-up evaluation after program completion.
  Interventions: Behavioral: Functional Exercise
- Control (Sham Comparator): Participants in the control group will receive weekly health newsletters and will not get any suggestions or encouragement to do exercise from the research team. A staff member will call the control group participants weekly to document any new exercise programs from usual community services. At this stage, participants will not be excluded from the study if they join an exercise program, but we will document what kind of exercise they are conducting. Trained raters will administer at post-tests and two follow-ups.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Functional Exercise — Treatment group will receive the 12-week STEP by a trained interventionist. During the intervention period, an occupational therapist will help the participant to learn the STEP exercise and principles and help the older adults to be more independent on functional exercising.
  Arms: Treatment
Behavioral: Education — In the education group, participant will receive weekly health newsletters containing general health aging materials. A staff member will call the control group participants weekly to document any new exercise programs from usual community services.
  Arms: Control

SUMMARY:
Sarcopenia is one of the major causes of functional decline and negative health outcomes among older adults. Prominent evidence suggests exercise interventions can reverse sarcopenia. However, past studies mainly focus on structured exercise programs, automatically excluding many older adults who are not motivated and lack the time/resources to conduct the structural exercise. Therefore, we propose to examine the effect of the Sarcopenia Translation functional Exercise Program (the STEP program) on community-dwelling older adults. The STEP is a functional exercise program designed to address low motivation and other time/resources barriers for rapid translation in community settings. The 12-week STEP program teaches older adults to apply functional exercise activities incorporating resistant training principles in their daily routines.

With a dual focus apriori in assessing clinical effectiveness and potential implementation strategies for future community implementations, we will conduct a single-blind randomized control trial among 60 community-dwelling older adults at risk or with sarcopenia. The study's purposes are threefold: (1) to assess the effect of the functional exercise intervention compared to usual care on primary outcomes of sarcopenia (muscle strength, muscle mass, and physical function); (2) to assess the long-term effects of the functional exercise intervention on primary outcomes of sarcopenia; (3) explore potential implementation strategies for rapid community implementation including development of a communityappropriate protocol for tracking long-term effects such as metabolomic biomarkers. This study aims to develop an effective functional exercise program as an alternative to structured exercise programs. Additionally, the goal is to accelerate the translation of the functional exercise program for older adults at risk or with sarcopenia in real-world settings.

ELIGIBILITY:
Inclusion Criteria:

1. age 65 or older
2. reside in northern Taiwan
3. at risk of /with sarcopenia determined by AWGS diagnostic guidelines

Exclusion Criteria:

1. meets physical activity guidelines for older adults: conduct at least 150 minutes of moderate-intensity activity or 75 minutes of vigorous-intensity activity weekly
2. needs 24-hour resistance for the activity of daily living activities
3. has severe knee or back pain
4. severely impaired mobility or wheelchair bounded (ruling out possible secondary sarcopenia patients)
5. unstable cardiac conditions such as ventricular dysrhythmias, pulmonary edema, or other musculoskeletal conditions
6. impaired cognition (Mini-Mental State Examination [MMSE] score < 24, or <17 for participants with lower education level)
7. has a metal clip, implant, or pacemaker

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of skeletal muscle strength in 12 weeks and 3 and 6 month follow-ups | From baseline to 6 month follow-up
  Using a handheld dynamometer (MicroFET2, MMT) to measure the maximal isometric knee strength of the dominant leg with a standardized protocol.
Change of muscle mass in 12 weeks and 3 and 6 month follow-ups | From baseline to 6 month follow-up
  Skeletal muscle mass will be measured by a portable Bio-impedance analysis (BIA) instrument at 50hz (Yida muscle mass and strength analyzer; YD01A), which had preliminary valid data for Taiwanese older adults and can be easily carried to community settings.
Change of physical performance in 12 weeks and 3 and 6 month follow-ups | From baseline to 6 month follow-up
  The Short Physical Performance Battery (SPPB) is an assessment of lower extremity function with three subtests: (1) standing balance, (2) four-meter gait speed, and (3) five repetitions of sit-to-stand motion.
The Reach, Adoption, Adherence and Fidelity of this research. | From baseline to 6 month follow-up
  Reach includes recruitment and retention rates. Adoption will be surveyed among participants and service networks at post-test. Adherence will be measured by the average number of activities recorded in the STEP activity planner. Fidelity is defined as treatment delivery, treatment receipt, and treatment enactment.

SECONDARY OUTCOMES:
Change of exercise habit in 12 weeks and 3 and 6 month follow-ups | From baseline to 6 month follow-up
  Self-Reported Habit Index (SRHI), a self-rated assessment, which incorporates constructs such as habit strength, frequency, relevance to self-identity, and automaticity. Higher scores indicate that behavior is more strongly habitual.
Change of sedentary time in 12 weeks and 3 and 6 month follow-ups | From baseline to 6 month follow-up
  Participants will wear an ActiGraph accelerometer over the right hip on an elasticized belt for seven days after the consent visit. Participants will be asked to wear the accelerometer throughout the day except swimming, showering, or bathing.
Change of quality of life in 12 weeks and 3 and 6 month follow-ups | From baseline to 6 month follow-up
  The Chinese The World Health Organization Quality of Life-Brief assessment (WHOQoL-BREF) is a validated measure that assesses physical, psychological, social relationships, and environmental quality of life.

CONTACTS AND LOCATIONS:
Locations (7):
- Taiwan (7):
  - Pei Ai holistic care association, New Taipei City
  - Silver Care Association, New Taipei City
  - Chinese e-touch community service association, Taoyuan District
  - Family Caregiver Care Association, Taoyuan District
  - Social Service Care Association (Guishan District), Taoyuan District
  - Waishe community association, Taoyuan District
  - Zhongshan community association, Taoyuan District

IPD SHARING:
Plan to Share IPD: No